CLINICAL TRIAL: NCT06238817
Title: A Phase 3b, Double-Blind, Multicenter, Randomized, Vehicle-Controlled, Efficacy, and Safety Study of Ruxolitinib Cream in Adults With Moderate Atopic Dermatitis
Brief Title: A Study to Evaluate the Efficacy, and Safety Study of Ruxolitinib Cream in Adults With Moderate Atopic Dermatitis
Acronym: TRuE-AD4
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: INCB18424-326; 2023-505433-27-00 (Registry Identifier: EU CT Number)
Record Dates: First submitted 2024-01-25; First posted 2024-02-02 (Actual); Last update posted 2025-10-28 (Actual); Status verified 2025-10

CONDITIONS: Atopic Dermatitis
Keywords: Atopic dermatitis; pruritus; eczema; topical therapy; JAK inhibitor
MeSH Terms: conditions — Dermatitis, Atopic; Pruritus; Eczema

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- VC Period: Ruxolitinib 1.5% Cream BID (Experimental): Participants received ruxolitinib 1.5% cream, applied topically to the affected areas as a thin film twice daily (BID) from Day 1 to Week 8 during the Vehicle Control (VC) Period. Participants applied cream BID to areas identified at Baseline even if the areas improved.
  Interventions: Drug: Ruxolitinib Cream
- VC Period: Vehicle Cream BID (Placebo Comparator): Participants received vehicle cream, applied topically to the affected areas as a thin film twice daily (BID) from Day 1 to Week 8 during the VC Period. Participants applied cream BID to areas identified at Baseline even if the areas improved.
  Interventions: Drug: Vehicle Cream
- VC Extension Period/Escape Arm: Ruxolitinib 1.5% Cream BID (Experimental): Participants who applied ruxolitinib 1.5% cream during VC Period, continued applying ruxolitinib 1.5% cream topically to the affected areas as a thin film BID from Week 8 to 24 during the Vehicle Control Extension (VCE) Period. Participants stopped treatment 3 days after lesions disappeared and restarted at the first sign of recurrence.
  Interventions: Drug: Ruxolitinib Cream
- VC Extension Period/Escape Arm: Vehicle Cream BID (Placebo Comparator): Participants who applied vehicle cream during the VC Period, continued applying vehicle cream as a thin film twice daily (BID) from Weeks 8 to 24 during the VCE Period. Participants applied cream BID to areas identified at Baseline even if the areas improved. Participants will be eligible to enter the ruxolitinib 1.5% cream open-label escape arm as defined in the protocol.
  Interventions: Drug: Vehicle Cream
- VC Extension Period: Ruxolitinib 1.5% cream open-label escape arm (Experimental): Participants received ruxolitinib 1.5% cream, applied topically to the affected areas as a thin film twice daily (BID) during the VCE Period. Participants applied cream BID to areas identified at Baseline even if the areas improved.
  Interventions: Drug: Ruxolitinib Cream

INTERVENTIONS:
Drug: Ruxolitinib Cream — Ruxolitinib cream applied topically to the affected area as a thin film twice daily.
  Other Names: INCB018424 Phosphate Cream
  Arms: VC Extension Period/Escape Arm: Ruxolitinib 1.5% Cream BID; VC Extension Period: Ruxolitinib 1.5% cream open-label escape arm; VC Period: Ruxolitinib 1.5% Cream BID
Drug: Vehicle Cream — Matching vehicle cream applied topically to the affected area as a thin film twice daily.
  Arms: VC Extension Period/Escape Arm: Vehicle Cream BID; VC Period: Vehicle Cream BID

SUMMARY:
This study is being conducted to establish the efficacy of ruxolitinib cream in participants with moderate AD who had an inadequate response to, or are intolerant to, or contraindicated to topical corticosteroid (TCS)s and topical calcineurin inhibitor (TCI)s.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged ≥ 18 years at screening (Note: Legal adult age for Korea is ≥ 19 years).
* Diagnosis of AD as defined by the Hanifin and Rajka (1980) criteria.
* AD duration of at least 2 years.
* IGA score of 3 at screening and Day 1.
* EASI score > 7 at screening and Day 1.
* Itch NRS score ≥ 4 at Day 1, defined as the average of the 7 days directly before Day 1, with Itch NRS values available for at least 4 of the 7 days.
* %BSA (excluding the scalp) with AD involvement of at least 10% and up to 20% at screening and Day 1.
* DLQI score > 10 at screening and Day 1.
* Documented recent history (within 12 months before the screening visit) of inadequate response, intolerance, or contraindication to TCSs and TCIs.
* Agree to discontinue all agents used to treat AD from screening through the final follow up visit, except as outlined in the protocol.
* Willingness to avoid pregnancy or fathering children based on the criteria as outlined in the protocol.

Exclusion Criteria:

* Unstable course of AD (spontaneously improving or rapidly deteriorating) as determined by the investigator in the 4 weeks prior to Day 1.
* Concurrent conditions and history of other diseases as follows:

  * Immunocompromised (eg, lymphoma, acquired immunodeficiency syndrome, Wiskott-Aldrich syndrome).
  * Chronic or acute infection requiring treatment with systemic antibiotics, antivirals, antiparasitics, antiprotozoals, or antifungals within 2 weeks before Day 1.
  * Active acute bacterial, fungal, or viral skin infection (eg, herpes simplex, herpes zoster, chickenpox) within 1 week before Day 1.
  * Any other concomitant skin disorder (eg, generalized erythroderma, such as Netherton syndrome), pigmentation, or extensive scarring that, in the opinion of the investigator, may interfere with the evaluation of AD lesions or compromise participant safety.
  * Presence of AD lesions only on the hands or feet without prior history of involvement of other classic areas of involvement such as the face or the flexural folds.
  * Other types of eczema within the 6 months prior to screening. Note: Seborrheic dermatitis on the scalp is allowed, as the scalp will not be treated with study cream.
  * Current or history of hepatitis B or C virus infection.
* Any serious illness or medical, physical, or psychiatric condition(s) that, in the investigator's opinion, would interfere with full participation in the study, including administration of study cream and attending required study visits; pose a significant risk to the participant; or interfere with interpretation of study data.
* Any of the following clinical laboratory test results at screening:

  * Hemoglobin < 10 g/dL.
  * Liver function tests:

    * AST or ALT ≥ 2 × ULN.
    * Alkaline phosphatase > 1.5 × ULN.
    * Bilirubin > 1.5 × ULN (isolated bilirubin > 1.5 × ULN is acceptable if bilirubin is fractionated and direct bilirubin < 35%) with the exception of Gilbert's disease.
  * Estimated glomerular filtration rate < 30 mL/min/1.73 m2 (using the Chronic Kidney Disease Epidemiology Collaboration equation).
  * Positive serology test results for HIV antibody.
  * Any other clinically significant laboratory result that, in the opinion of the investigator, poses a significant risk to the participant.
* Use of any of the following treatments within the indicated washout period before Day 1:

  * 5 half-lives or 12 weeks, whichever is longer: biologic agents. For biologic agents with washout periods longer than 12 weeks (eg, rituximab), consult the medical monitor.
  * 4 weeks: systemic corticosteroids or adrenocorticotropic hormone analogs, cyclosporine, methotrexate, azathioprine, or other systemic immunosuppressive (eg, JAK inhibitors) or immunomodulating agents (eg, mycophenolate or tacrolimus).
  * 2 weeks or 5 half-lives, whichever is longer - strong systemic CYP3A4 inhibitors.
  * 2 weeks: immunizations with live-attenuated vaccines; sedating antihistamines unless on a long-term stable regimen (nonsedating antihistamines are permitted).

Note: COVID-19 vaccination is allowed.

• 1 week: use of other topical treatments for AD, other than bland emollients (eg, Aveeno creams, ointments, sprays, soap substitutes), such as antipruritics (eg, doxepin cream), corticosteroids, calcineurin inhibitors, PDE4 inhibitors, coal tar (shampoo), antibiotics, or antibacterial cleansing body wash/soap.

Note: Diluted sodium hypochlorite "bleach" baths are allowed as long as they do not exceed 2 baths per week and their frequency remains the same throughout the study.

* History of treatment failure with any systemic or topical JAK inhibitor (eg, ruxolitinib, tofacitinib, baricitinib, abrocitinib, upadacitinib) for AD or any other inflammatory condition.
* Ultraviolet light therapy or prolonged exposure to natural or artificial sources of UV radiation (eg, sunlight or tanning booth) within 2 weeks prior to the baseline visit and/or intention to have such exposure during the study that is thought by the investigator to potentially impact the participant's AD.
* Current treatment or treatment within 30 days or 5 half-lives (whichever is longer) before baseline with another investigational medication or current enrollment in another investigational drug protocol.
* In the opinion of the investigator, are unable or unlikely to comply with the administration schedule, study evaluations, and procedures (eg, eDiary compliance).

Other protocol-defined Inclusion/Exclusion Criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 241 (Actual)
Dates: Start 2024-04-26 (Actual); Primary Completion 2025-05-21 (Actual); Study Completion 2025-10-17 (Actual)

PRIMARY OUTCOMES:
VC Period: Proportion of participants who achieved Eczema Area and Severity Index 75 (EASI75) | Baseline to Week 8
  Defined as ≥ 75% improvement in Eczema Area and Severity Index (EASI) score.
VC Period: Proportion of participants who achieved Investigator's Global Assessment Treatment Success (IGA-TS) | Baseline to Week 8
  Defined as Investigator's Global Assessment (IGA) score of 0 or 1 with ≥ 2 grade improvement from baseline.

SECONDARY OUTCOMES:
VC Period: Proportion of participants with a ≥ 4-point improvement in Itch Numeric Rating Scale (NRS) score (ITCH4) | Baseline to Week 8
  ITCH4 is defined as achieving ≥ 4-point improvement in Itch NRS score.
VC Period: Proportion of participants with a ≥ 4-point improvement in Itch Numeric Rating Scale (NRS) score (ITCH4) | Baseline to Day 7
  ITCH4 is defined as achieving ≥ 4-point improvement in Itch NRS score.
VC Period: Proportion of participants with a ≥ 4-point improvement in Itch Numeric Rating Scale (NRS) score (ITCH4) | Baseline to Day 3
  ITCH4 is defined as achieving ≥ 4-point improvement in Itch NRS score.
VC Period: Proportion of participants with a ≥ 4-point improvement in Itch Numeric Rating Scale (NRS) score (ITCH4) | Baseline to Day 2
  ITCH4 is defined as achieving ≥ 4-point improvement in Itch NRS score.
VC Period: Number of Treatment Emergent Adverse Events (TEAEs) | Up to Week 24, followed by 30 days follow-up
  An AE is any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug-related. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of study treatment. A SAE is defined as any untoward medical occurrence that, at any dose results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect or an important medical event may be considered serious when, based on appropriate medical judgment, the event may jeopardize the participant and may require medical or surgical intervention to prevent one of the outcomes listed above. A TEAE or treatment emergent SAE is any AE or SAE either reported for first time or worsening of a pre-existing event after first dose of study drug.
VC Period: Proportion of participants who achieved Eczema Area and Severity Index 75 (EASI75) | Baseline to Weeks 2 and 4
  Defined as ≥ 75% improvement in Eczema Area and Severity Index (EASI) score.
VC Period: Proportion of participants who achieved Investigator's Global Assessment - Treatment Success (IGA-TS) | Baseline to Weeks 2 and 4
  Defined as Investigator's Global Assessment (IGA) score of 0 or 1 with ≥ 2 grade improvement from baseline.
VC Period: Proportion of participants with a ≥ 4-point improvement in Itch Numeric Rating Scale (NRS) score (ITCH4) | Baseline to Weeks 2 and 4
  ITCH4 is defined as achieving ≥ 4-point improvement in Itch NRS score.
VC Period: Time to achieve a ≥ 4-point improvement in Itch Numeric Rating Scale (NRS) score (ITCH4) | Baseline to Week 8
  ITCH4 is defined as achieving ≥ 4-point improvement in Itch NRS score.
VC Period: Time to achieve ≥ 2-point improvement from in Itch Numeric Rating Scale (NRS) score (ITCH2) | Baseline to Week 8
  ITCH2 is defined as achieving ≥ 2-point improvement from baseline in Itch NRS score.
VC Period: Change from baseline (pre-study cream application) in current Itch NRS score at 5, 15, 30, 45, and 60 minutes and 2, 4, and 6 hours post-initial dose on Day 1. | Baseline to Day 1
VC Period: Proportion of participants achieving at least a 2-point decrease from baseline in current Itch NRS score at 5, 15, 30, 45, and 60 minutes and 2, 4, and 6 hours post-initial dose on Day 1. | Baseline to Day 1
VC Period: Proportion of participants achieving at least a 4-point decrease from baseline in current Itch NRS score at 5, 15, 30, 45, and 60 minutes and 2, 4, and 6 hours post-initial dose on Day 1. | Baseline to Day 1
VC and VCE Periods: Proportion of participants who achieved EASI50 | Baseline to Weeks 2, 4, 8, 12, 16, 20 and 24
  Defined as ≥ 50% improvement in Eczema Area and Severity Index (EASI) score.
VC and VCE Periods: Proportion of participants who achieved EASI90 | Baseline to Weeks 2, 4, 8, 12, 16, 20 and 24
  Defined as ≥ 90% improvement in Eczema Area and Severity Index (EASI) score.
VC and VCE Periods: Proportion of participants achieving both EASI75 and IGA-TS | Baseline to Weeks 2, 4, 8, 12, 16, 20 and 24
  Defined as ≥ 75% improvement in Eczema Area and Severity Index (EASI) score and IGA score of 0 or 1 with ≥ 2 grade improvement from baseline.
VC and VCE Periods: Change from Baseline in Atopic Dermatitis Afflicted Percentage of Body Surface Area (%BSA) | Baseline to Weeks 2, 4, 8, 12, 16, 20 and 24
  A negative change from Baseline indicates improvement.
VC and VCE Periods: Change from baseline in EASI score | Baseline to Weeks 2, 4, 8, 12, 16, 20 and 24
  A negative change from Baseline indicates improvement.
VC and VCE Periods: Change from baseline in SCORAD score | Baseline to Weeks 2, 4, 8, 12, 16, 20 and 24
  SCORing Atopic Dermatitis - tool used to assess extent and severity (intensity) of eczema.
VC and VCE Periods: Change from baseline in Itch NRS score | Baseline to Weeks 2, 4, 8, 12, 16, 20 and 24
  The Itch NRS is an instrument for measurement of itch intensity and participant will rate the intensity of their itch on an 11-point scale ranging from 0 (no itch) to 10 (worst itch imaginable).
VC and VCE Periods: Change from baseline in Skin Pain NRS score | Baseline to Weeks 2, 4, 8, 12, 16, 20 and 24
  The Skin Pain NRS is a daily participant-reported measure (24-hour or 7-day recall) of the worst level of pain intensity from 0 (no pain) to 10 (worst pain imaginable.
VCE Period: Time to open-label escape arm | Baseline to Week 24
  Defined as not achieving 50% improvement in EASI score from baseline at 2 consecutive visits at least 1 week apart.
VC and VCE Periods: Proportion of participants concurrently meeting all of the following criteria: IGA score ≥ 3, EASI score ≥ 16, Itch NRS score ≥ 4, BSA ≥ 10%, and DLQI score > 10 | Baseline to Weeks 2, 4, 8, 12, 16, 20 and 24
VC and VCE Periods: Time to concurrently meeting all of the following criteria: IGA score ≥ 3, EASI score ≥ 16, Itch NRS score ≥ 4, BSA ≥ 10%, and DLQI score > 10 | Baseline to Week 24
VC Period: Proportion of participants who experience a relapse after study treatment discontinuation | Week 24 to Follow-up (30 days)
  Defined as proportion of participants among EASI75 responders who are on study treatment at Week 24 who meet relapse criteria [loss of EASI50 from baseline] at the safety follow-up visit.
VCE period: Time to first re-treatment | Week 8 to Week 24
VCE Period: Proportion of time off study treatment due to lesion clearance | Week 8 to Week 24
VCE period: Proportion of time on study treatment | Week 8 to Week 24
VC and VCE Periods: Proportion of participants who achieve ≥ 4-point improvement in DLQI from baseline | Baseline to Weeks 2, 4, 8, 12, 16, 20 and 24
  The DLQI is a 10-question validated questionnaire to measure how much the skin problem has affected the participant over the previous 7 days. The participant will answer the questionnaire with either (1) very much, (2) a lot, (3) a little, or (4) not at all. A negative change from Baseline indicates less impact of the skin problem on participant's life.
VC and VCE Periods: Change From Baseline in Dermatology Life Quality Index (DLQI) Score | Baseline to Weeks 2, 4, 8, 12, 16, 20 and 24
  The DLQI is a 10-question validated questionnaire to measure how much the skin problem has affected the participant over the previous 7 days. The participant will answer the questionnaire with either (1) very much, (2) a lot, (3) a little, or (4) not at all. A negative change from Baseline indicates less impact of the skin problem on participant's life.
VC and VCE Periods: Change From Baseline in Patient-Oriented Eczema Measure (POEM) Score | Baseline to Weeks 2, 4, 8, 12, 16, 20 and 24
  The POEM is a 7-question quality-of-life assessment that asks how many days the participant has been bothered by various aspects of their skin condition during the past 7 days. A negative change from Baseline indicates improvement.
VC and VCE Periods: Change From Baseline in EuroQuality of Life Five Dimensions (EQ-5D-5L) Visual Analogue Scale (VAS) Score | Baseline to Weeks 2, 4, 8, 12, 16, 20 and 24
  he EQ-5D-5L questionnaire is a standardized, validated instrument for use as a measure of health outcome. The descriptive system comprises 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has 5 levels: Level 1 = no problems, Level 2 = slight problems, Level 3 = moderate problems, Level 4 = severe problems, and Level 5 = extreme problems.
VC and VCE Periods: Change from baseline in the HADS scores | Baseline to Weeks 2, 4, 8, 12, 16, 20 and 24
  The Hospital Anxiety and Depression Scale (HADS) is a 14-item questionnaire to be completed by tablet; the questionnaire assesses the levels of anxiety and depression a person is currently experiencing. There are 7 questions each for measuring anxiety and for measuring depression, with 4 possible responses to each question (responses are scored as 0, 1, 2, or 3). Separate scores are calculated for anxiety and depression. The recall period will be the past 7 days for both the VC and VCE periods.
VC and VCE Periods: Change from baseline in PROMIS Short Form - Sleep-Related Impairment (8a) 24-Hour Recall Score | Baseline to Weeks 2, 4, 8, 12, 16, 20 and 24
  The Patient-Reported Outcomes Measurement Information System (PROMIS) Short Form - Sleep-Related Impairment (8a) questionnaire assesses participant's self-reported perceptions of alertness, sleepiness, and tiredness during usual waking hours and the perceived functional impairments during wakefulness associated with sleep problems or impaired alertness. The questionnaire is filled in the evening where each item asks the participant to rate the severity of the participant's sleep impairment. It has 8 simple questions with a 5-point scale with a range in score from 8 to 40, with higher scores indicating greater severity of sleep-related impairment. A negative change from Baseline indicates improvement.
VC and VCE Period: Change From Baseline in PROMIS Short Form - Sleep Disturbance (8b) 7-Day Recall Score | Baseline to Weeks 2, 4, 8, 12, 16, 20 and 24
  The PROMIS Short Form - Sleep Disturbance (8b) questionnaire assesses participant's self-reported perceptions of sleep quality, sleep depth, and restoration associated with sleep. This questionnaire is completed in the morning by the participant where each item asks the participant to rate the severity of the participant's sleep disturbance. It is a 5-point scale with a range in score from 8 to 40, with higher scores indicating greater severity of sleep disturbance. A negative change from Baseline indicates improvement.
VC and VCE Periods: Change from baseline score in Work Productivity and Activity Impairment - Atopic Dermatitis (WPAI-AD) | Baseline to Week 8 and Week 24
  The WPAI-AD questionnaire is a validated 6-item instrument that measures the effect of overall health and specific symptoms on productivity at work and regular activities outside of it during the past 7 days.

CONTACTS AND LOCATIONS:
Overall Officials: Incyte Medical Monitor, Study Director — Incyte Corporation
Locations (94):
- United States (18):
  - Lynn Institute of the Ozarks, Little Rock, Arkansas
  - First Oc Dermatology, Fountain Valley, California
  - Center For Dermatology Cosmetic and Laser Surgery, Fremont, California
  - Medderm Associates, Inc, San Diego, California
  - Encore Medical Research, Llc Hollywood, Hollywood, Florida
  - Entrust Clinical Research, Miami, Florida
  - Lane Dermatology and Dermatologic Surgery, Columbus, Georgia
  - Marietta Dermatology the Skin Cancer Center Marietta, Marietta, Georgia
  - Arlington Dermatology, Rolling Meadows, Illinois
  - Northshore University Healthsystem, Skokie, Illinois
  - Oakland Hills Dermatology Pc, Auburn Hills, Michigan
  - Revival Research Institute, Llc Troy, Troy, Michigan
  - Best Skin Research, Camp Hill, Pennsylvania
  - International Clinical Research Tennessee Llc, Murfreesboro, Tennessee
  - Center For Clinical Studies Webster, Houston, Texas
  - Texas Dermatology Research Center, Plano, Texas
  - Rainey and Finklea Dermatology, San Antonio, Texas
  - North Sound Dermatology, Mill Creek, Washington
- Australia (6):
  - Premier Specialists Pty Ltd, Kogarah, New South Wales
  - Australian Clinical Research Network, Maroubra, New South Wales
  - Veracity Clinical Research, Woolloongabba, Queensland
  - Clinical Trials Sa, Campbelltown, South Australia
  - Skin Health Institute Inc., Carlton, Victoria
  - Paratus Clinical Research, Woden, Phillip
- Belgium (6):
  - Ulb Hospital Erasme, Brussels
  - Cliniques Universitaires Ucl Saint-Luc, Brussels
  - Universitair Ziekenhuis Antwerpen (Uza), Edegem
  - Universitair Ziekenhuis Gent (Uz Gent), Ghent
  - Grand Hopital de Charleroi, Gilly
  - Dermatologie Handelskaai, Kortrijk
- Bulgaria (7):
  - Mhat Dr. Tota Venkova Ad, Gabrovo
  - Medical Center Medconsult Pleven Ood, Pleven
  - Ambulatory For Specialized Medical Help - Skin and Venereal Diseases, Sofia
  - Dcc 'Alexandrovska', Eood, Sofia
  - Medical Center Hera Eood, Sofia
  - Diagnostic Consultative Center Xxviii, Sofia
  - Medical Center Assoc. Prof. Vasilev, Sofia
- Canada (8):
  - Dermatology Research Institute Inc., Calgary, Alberta
  - Dr. Chih-Ho Hong Medical Inc., Surrey, British Columbia
  - Wiseman Dermatology Research Inc, Winnipeg, Manitoba
  - Dr. Irina Turchin Pc Inc., Fredericton, New Brunswick
  - Lynderm Research Inc, Markham, Ontario
  - Skin Centre For Dermatology, Peterborough, Ontario
  - Centre de Recherche Dermatologique Du Quebec Metropolitain, Québec, Quebec
  - Skincare Studio Dermatology Centre, St. John's
- France (5):
  - Ghicl - Hôpital Saint-Vincent de Paul, Lille
  - Centre Hospitalier Universitaire de Nantes (Chu de Nantes) - Hotel-Dieu, Nantes
  - Hospices Civils de Lyon Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Chu de Rouen - Hospital Charles Nicolle, Rouen
  - University Hospital of Saint Etienne, Saint-Etienne
- Germany (5):
  - Universitaetsklinikum Augsburg Sued, Augsburg
  - Fachklinik Bad Bentheim Dermatologie, Bad Bentheim
  - Praxis Fuer Haut- Und Geschlechtskrankheiten Dr. Med. Thomas Wildfeuer Und Partner, Berlin
  - Universitatsklinikum Munster, Münster
  - Dermatologie Potsdam Mvz Gmbh, Potsdam
- Hungary (5):
  - Clinexpert Kft., Budapest
  - Obudai Egeszsegugyi Centrum Kft., Budapest
  - Semmelweis Egyetem, Budapest
  - Debreceni Egyetem Klinikai Kozpon Belgyogy Klinika, Debrecen
  - Szegedi Tudomanyegyetem Aok Szent-Gyorgyi Albert Klinikai Kozpont, Szeged
- Italy (5):
  - Fondazione Irccs Ca Granda Ospedale Maggiore, Milan
  - Azienda Ospedaliera Universitaria Federico Ii, Napoli
  - Universita Degli Studi Della Campania Luigi Vanvitelli, Napoli
  - Fondazione Policlinico Universitario Agostino Gemelli Irccs, Rome
  - Irccs Istituto Clinico Humanitas, Rozzano
- Netherlands (3):
  - Bravis Ziekenhuis, Bergen op Zoom
  - Amphia Ziekenhuis, Molengracht, Breda
  - Universitair Medisch Centrum Groningen, Groningen
- Poland (11):
  - Centrum Badan Klinicznych Pi-House Sp. Z O.O., Gdansk
  - Centrum Medyczne Pratia Katowice, Katowice
  - Centrum Medyczne All-Med, Krakow
  - Pratia McM Krakow, Krakow
  - Santa Sp. Z O.O. Santa Familia Ptg Lodz, Lodz
  - Etg Lublin, Lublin
  - Solumed Centrum Medyczne, Poznan
  - Twoja Przychodnia - Szczecinskie Centrum Medyczne, Szczecin
  - Centrum Medyczne Evimed, Warsaw
  - Klinika Ambroziak Dermatologia, Warsaw
  - Dermmedica Sp. Z O.O., Wroclaw
- Spain (6):
  - Ceim Hospital Universitari Germans Trias I Pujol, Badalona
  - Hospital de La Santa Creu I Sant Pau, Barcelona
  - Hospital Infanta Leonor, Madrid
  - Hospital Universitario de La Paz, Madrid
  - Hospital de Manises, Manises
  - Hospital Marina Baixa, Villajoyosa
- Switzerland (4):
  - Universitatsspital Basel, Basel
  - Inselspital Universitatsklinik Fur Medizinische Onkologie, Bern
  - Dermatology & Skin Care Clinic, Buochs
  - Universitatsspital Zurich, Zurich
- United Kingdom (5):
  - West Middlesex University Hospital, Isleworth
  - Guys Hospital, London
  - Northampton General Hospital, Northampton
  - University Hospital Plymouth, Plymouth
  - Walsall Manor Hospital, Walsall

IPD SHARING:
Plan to Share IPD: Yes
Incyte shares data with qualified external researchers after a research proposal is submitted. These requests are reviewed and approved by a review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations. The trial data availability is according to the criteria and process described on https://www.incyte.com/our-company/compliance-and-transparency
Supporting Information: Study Protocol, SAP
Time Frame: Data will be shared after the primary publication or 2 years after the study has ended for market authorized products and indications
Access Criteria: Data from eligible studies will be shared with qualified researchers according to the criteria and process described in the Data Sharing section of the www.incyteclinicaltrials.com website. For approved requests, the researchers will be granted access to anonymized data under the terms of a data sharing agreement.
URL: https://www.incyte.com/our-company/compliance-and-transparency

REFERENCES:
- See also: A study to evaluate the Efficacy, and Safety Study of Ruxolitinib Cream in Adults With Moderate Atopic Dermatitis — https://www.incyteclinicaltrials.com/study/?id=INCB18424-326&SearchTerm=INCB18424-326&Latitude=&Longitude=&LocationName=&conditions=&Status=&phases=&AgeRanges=&gender=&StudyTypes=&AttachmentTypes=&MileRadius=100&PageIndex=0&PageSize=10&SortField=&SortOrder=&hasResults=